CLINICAL TRIAL: NCT03136900
Title: Controlled, Randomized, Double-blind, Monocentric Clinical Study Evaluating the Impact on the Nitrogen Balance, Autonomy, Safety and Tolerance of Enteral Diets Made of Nutrilon Without Lactose® Fortified by Concentration Versus by Maltodextrin and Oil Supplementation, After Surgery for Congenital Heart Disease, in Children Aged Zero to Two Years Old
Brief Title: Impact on the Nitrogen Balance, Autonomy, Safety and Tolerance of Enteral Diets Made of With Nutrilon Without Lactose® Fortified by Concentration Versus by Maltodextrin and Oil Supplementation,After Surgery for Congenital Heart Disease, in Infants.
Acronym: DIETCHIRCARD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recuitment to slow
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: P2017/PICU/DIETCHIRCARD
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Congenital Heart Disease in Children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Diet (Experimental): Enteral diet made of Nutrilon without lactose® fortified by concentration
  Interventions: Dietary Supplement: Nutrilon without lactose® fortified by concentration
- Control Diet (Active Comparator): Enteral diet made of Nutrilon without lactose® fortified by Maltodextrin and oil supplementation.
  Interventions: Dietary Supplement: Nutrilon without lactose® fortified by Maltodextrin and oil supplementation

INTERVENTIONS:
Dietary Supplement: Nutrilon without lactose® fortified by concentration — enteral diet with cow milk protein-based infant formula without lactose 20% in place of 14%
  Arms: Study Diet
Dietary Supplement: Nutrilon without lactose® fortified by Maltodextrin and oil supplementation — enteral diet with cow milk protein-based infant formula without lactose 14%
  Arms: Control Diet

SUMMARY:
An adequate nutritional support after a cardiac surgery enhances the morbidity and mortality.

After a cardiac surgery, the energy expenditure is estimated to be around 55 kcal/kg/d. The caloric intake is not the only important nutritional variable in PICU. The protein intake objective is around 1,5g/kg/d in order to reduce muscular catabolism.

The aim of this study is to compare the impact of an isocaloric enteral diet, either fortified by milk concentration (in order to increase the protein intake) or by a supplement of maltodextrin and oil in children from 0 to 2 years, after surgery for congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Children from 0 to 2 years undergoing cardiac surgery (corrective or palliative) for congenital heart surgery, with or without extracorporeal circulation
* Expected stay of 5 days in PICU after surgery
* Expected need of invasive ventilation for 48h after surgery
* Expected need for enteral feeding during 5 days.
* Obtaining the informed consent of the child's legal guardian after being informed of the goals, benefits and potential risks of this study

Exclusion Criteria:

* Medical indications for specific diet
* ECMO
* Dialysis

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
positive nitrogen balance | Day 5 post operative

SECONDARY OUTCOMES:
duration of enteral feeding | up to 120 days post operative
  duration in hour
duration of invasive or non-invasive ventilatory support | up to 120 days post operative
  duration in hour
length of hospital stay in intensive care unit | up to 120 days post operative
  duration in hour
length of hospital stay in hospital | up to 120 days post operative
  duration in hour

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No